CLINICAL TRIAL: NCT06065046
Title: A Randomized Control Trial of Baricitinib Administration in Patients With Moderate and Severe Traumatic Intracerebral Hemorrhage/Contusions
Brief Title: Baricitinib for Moderate and Severe Traumatic Intracerebral Hemorrhage/Contusions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Qianxian People's Hospital (Unknown); Chongqing Hospital of PAP (Unknown); Weinan Central Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); the 987th Hospital of Chinese People's Liberation Army Joint Logistic Support Force (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDSJWK-TBI-Baritinib
Record Dates: First submitted 2023-07-04; First posted 2023-10-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic intracerebral Hemorrhage; traumatic intracerebral Contusions; baricitinib; Janus kinase inhibitor; neuro-inflammatory responses
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage, Traumatic | interventions — baricitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Participants will receive standard treatment and care according to the current management guidelines for traumatic brain injury, e.g. the guideline made by U.S. Brain Trauma Foundation (BTF)
  Interventions: Other: Standard treatment
- Baricitinib group (Experimental): Besides receiving standard treatment and care, baricitinib will be administrated orally (or crushed for nasogastric tube delivery) and given daily at the dosage of 4mg, for consecutive 14 days after patients' brain injury.
  Interventions: Drug: Baricitinib 4 MG

INTERVENTIONS:
Drug: Baricitinib 4 MG — Baricitinib with be be administrated orally (or crushed for nasogastric tube delivery) and given daily at the dosage of 4mg for consecutive 14 days
  Other Names: Baricitinib
  Arms: Baricitinib group
Other: Standard treatment — Patients will receive standard treatment and care according to the current management guidelines for traumatic brain injury.
  Other Names: Blank control
  Arms: Control group

SUMMARY:
The purpose of the present study is to study the effect of baricitinib administration on outcome of participants with moderate and severe traumatic intracerebral hemorrhage/contusions. A multi-center randomized control trial will be conducted. Participants with a radiological diagnosis of traumatic intracerebral hemorrhage/contusions and an initial GCS score of 5-12 will be screened and enrolled in the first 24 hours after traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains one of the biggest public health problems and represents a major cause of death or severe disability in young people and adults. Previous studies have confirmed that an infammatory response occurs directly after TBI, which contribute to the development of cerebral edema and swelling, a breakdown of the blood-brain barrier, and delayed neuronal cell death, thus application of agents with anti-infammatory actions may be promising to improve the functional outcomes for TBI patients. Activated Janus kinases (JAKs) play pivotal roles in intracellular signaling from cell-surface receptors for multiple cytokines implicated in the pathologic processes of TBI, selective JAK1 and JAK2 inhibitors (AG490 and abroctinib) have been shown to reduce the brain edema and improve neurological function for TBI rodents. Baricitinib, an orally available small molecule, provides reversible inhibition of JAK1 and JAK2 and has shown clinical efficacy in studies involving patients with rheumatoid arthritis, COVID-19 and alopecia areata, and was very safe for patients. Therefore, in the current study, a multicenter randomized control trial will be conducted to study the therapeutic efficacy of baricitinib for patients with moderate and severe traumatic intracerebral hemorrhage/contusions, comparing with the standard treatment only.The patients with the GCS scores of 5-12 will be enrolled according to the inclusive and exclusive criteria. The primary outcome is the Glasgow Outcome Scale at 180 days after brain trauma. And the secondary outcome including In-hospital mortality rate, and mortality rate at 90 days, 180 days after brain trauma; Glasgow Coma Scale at discharge; The Glasgow Outcome Scale at 90 days after brain trauma; The levels of serum inflammatory factors TNF-α、IFN-γ、IL-1β、IL-6、IL-8 at 2 to 7 days after brain trauma; Volume of edema around intracerebral hemorrhage/contusions at 2 to 7 days after brain trauma;The mean value of intracranial pressure at 2 to 7 days after brain trauma and The incidence of in-hospital pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years older and younger than 80 years old.
2. Definite history of traumatic brain injury.
3. Admission within≤24 hours after the traumatic brain injury.
4. CT scans demonstrate intracerebral hemorrhage/contusions with and without extracerebral hemorrhage (epi- and sub- dural hemorrhage)
5. GCS score of 5 or greater and no more than 12 at time of enrollment.
6. Closed head injury.
7. Admission without infections
8. Signed and dated informed consent by the subject, legally authorized representative, or surrogate obtained.

Exclusion Criteria:

1. Time of head injury cannot be reliably assessed.
2. Subjects is considered a candidate for immediate surgical intervention because of severe extracranial injury.
3. Open head injury.
4. Pregnancy or parturition within previous 30 days or active lactation.
5. Use of Janus kinase inhibitors (baricinitib,abroctinib, AG490 and etc.)
6. Pre-traumatic dementia or disability.
7. With severe liver, kidney disease, or malignancy, life expectancy is less than 14 days.
8. Severe pulmonary infection.
9. Severe or acute heart failure.
10. Severe infections within previous 30 days.
11. History of myocardial infarction.
12. Known sensitivity to baricinitib.
13. Severe decreases in neutrophil, lymphocyte and platelet counts, severe decrease in hemoglobin.
14. Severe liver and kidney dysfunction.
15. Currently participating in other interventional clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | up to 180 days
  Glasgow Outcome Scale at 180 days after brain trauma

SECONDARY OUTCOMES:
Mortality rate | up to 180 days
  In-hospital mortality rate, and mortality rate at 90 days, 180 days after brain trauma
Coma severity | up to 2 weeks
  Glasgow Coma Scale at baseline, and at discharge
Glasgow Outcome Scale | up to 90 days
  The Glasgow Outcome Scale at 90 days after brain trauma
Serum inflammatory factors | up to 7 days
  The levels of serum inflammatory factors TNF-α、IFN-γ、IL-1β、IL-6、IL-8 at 2 to 7days after brain trauma
Volume of edema around intracerebral hemorrhage/contusions | up to 7 days
  Volume of edema around intracerebral hemorrhage/contusions at 2 to 7days after brain trauma
Intracranial pressure | up to 7 days
  The mean value of intracranial pressure at 2 to 7 days after brain trauma
The incidence of pneumonia | up to 2 weeks
  The incidence of in-hospital pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, M.D,Ph.D, Study Chair — Tang-Du Hospital; Shunnan Ge, M.D,Ph.D, Study Director — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Begemann M, Leon M, van der Horn HJ, van der Naalt J, Sommer I. Drugs with anti-inflammatory effects to improve outcome of traumatic brain injury: a meta-analysis. Sci Rep. 2020 Sep 30;10(1):16179. doi: 10.1038/s41598-020-73227-5. PMID 32999392
- [Background] Jorgensen SCJ, Tse CLY, Burry L, Dresser LD. Baricitinib: A Review of Pharmacology, Safety, and Emerging Clinical Experience in COVID-19. Pharmacotherapy. 2020 Aug;40(8):843-856. doi: 10.1002/phar.2438. Epub 2020 Jul 27. PMID 32542785
- [Background] Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, Del Carmen Morales L, Reyes Gonzaga J, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich C, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka Y. Baricitinib versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2017 Feb 16;376(7):652-662. doi: 10.1056/NEJMoa1608345. PMID 28199814
- [Background] DU AL, Ji TL, Yang B, Cao JF, Zhang XG, Li Y, Pan S, Zhang B, Hu ZB, Zeng XW. Neuroprotective effect of AG490 in experimental traumatic brain injury of rats. Chin Med J (Engl). 2013;126(15):2934-7. PMID 23924471
- [Background] Li T, Li L, Peng R, Hao H, Zhang H, Gao Y, Wang C, Li F, Liu X, Chen F, Zhang S, Zhang J. Abrocitinib Attenuates Microglia-Mediated Neuroinflammation after Traumatic Brain Injury via Inhibiting the JAK1/STAT1/NF-kappaB Pathway. Cells. 2022 Nov 13;11(22):3588. doi: 10.3390/cells11223588. PMID 36429017
- [Background] Messenger A, Harries M. Baricitinib in Alopecia Areata. N Engl J Med. 2022 May 5;386(18):1751-1752. doi: 10.1056/NEJMe2203440. No abstract available. PMID 35507486
- [Background] Marconi VC, Ramanan AV, de Bono S, Kartman CE, Krishnan V, Liao R, Piruzeli MLB, Goldman JD, Alatorre-Alexander J, de Cassia Pellegrini R, Estrada V, Som M, Cardoso A, Chakladar S, Crowe B, Reis P, Zhang X, Adams DH, Ely EW; COV-BARRIER Study Group. Efficacy and safety of baricitinib for the treatment of hospitalised adults with COVID-19 (COV-BARRIER): a randomised, double-blind, parallel-group, placebo-controlled phase 3 trial. Lancet Respir Med. 2021 Dec;9(12):1407-1418. doi: 10.1016/S2213-2600(21)00331-3. Epub 2021 Sep 1. PMID 34480861